CLINICAL TRIAL: NCT01937585
Title: Evaluation of a Culturally Targeted, Personalized Mail-Home Brochure Directed to Partners of At-Risk Men to Facilitate Prostate Cancer Risk Assessment
Brief Title: Trial of Print Messages to Support the Role of Partners in Promoting Provider Discussions About Prostate Cancer Screening Among AA Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Knowledge Networks (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTMHB-DOD; W81XWH-06-1-0099 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2013-08-30; First posted 2013-09-09 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; partner; communication messages; monitoring style; AA men
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CDC brochure only condition (Active Comparator): Receipt of CDC brochure by female partners of African American men designed to provide African American men information and guidance concerning whether to undergo PSA and/or DRE screening for prostate cancer
  Interventions: Behavioral: CDC brochure only condition
- Partner and CDC brochure condition (Experimental): Receipt of a brochure designed for female partners of African American men designed to provide information about prostate cancer screening and strategies for influencing her mate to schedule a discussion with a health care provider about whether to undergo prostate cancer screening, in combination with receipt of the comparator brochure (CDC brochure for African American about prostate cancer screening).
  Interventions: Behavioral: Partner and CDC brochure condition

INTERVENTIONS:
Behavioral: Partner and CDC brochure condition — Receipt of a brochure designed for female partners of African American men designed to provide information about prostate cancer screening and strategies for influencing her mate to schedule a discussion with a health care provider about whether to undergo prostate cancer screening, in combination with receipt of the comparator brochure (CDC brochure for African American about prostate cancer screening).
  Arms: Partner and CDC brochure condition
Behavioral: CDC brochure only condition — Receipt of CDC brochure by female partners of African American men designed to provide African American men information and guidance concerning whether to undergo PSA and/or DRE screening for prostate cancer
  Arms: CDC brochure only condition

SUMMARY:
The purpose of this study is to determine whether female partners of African American men can promote initiation of a discussion with a healthcare provider about prostate cancer screening when the partner is supported by a print message designed to provide relevant information and strategies for her to use in this effort.

DETAILED DESCRIPTION:
Objective: Although AA men are at elevated risk for prostate cancer (Pca), medical guidelines do not present consistent screening recommendations for this group. However, all guidelines stress the need for screening decision making with a provider. This study evaluated the effectiveness of a brochure designed for the female partners of AA men, designed to help promote such discussion on the part of their mates. We also explored the effect of the partner's monitoring style (i.e., the extent to which the partner typically attends to health threats) on promoting discussion.

Methods: Female partners of AA men (N=231) were randomized to receive either a Pca screening CDC brochure for AA men, combined with a "partner" brochure containing strategies to promote men's initiation of a provider visit to discuss screening, or the CDC brochure only, and completed pre- and post-intervention surveys online.

Conclusions: High monitoring partners may be effective in influencing their AA mates to initiate provider discussion, particularly when tailored messaging is provided.

ELIGIBILITY:
Inclusion Criteria:

* U.S. female aged 18 and over, and having an AA male partner between the ages of 35 and 69 with no history of a Pca diagnosis

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Partner-reported actions of mate to initiate a provider visit to discuss prostate cancer screening | Two weeks post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne M Miller, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Sajid S, Kotwal AA, Dale W. Interventions to improve decision making and reduce racial and ethnic disparities in the management of prostate cancer: a systematic review. J Gen Intern Med. 2012 Aug;27(8):1068-78. doi: 10.1007/s11606-012-2086-5. PMID 22798216